CLINICAL TRIAL: NCT02635087
Title: microRNAs Tool for Stratifying Stage II Colon Cancer:a Perspective Study of Adjuvant Chemotherapy
Brief Title: microRNAs Tool for Stratifying Stage II Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wu Song, archiater, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2015[112]
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Colonic Neoplasms; Effects of Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will use the samples to make q-RT-PCR of our miRNA tool,then predict the patients as high risk one or not.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- high risk group: the miRNA tool predict this group of patients as "high risk"
  Interventions: Device: miRNA tool

INTERVENTIONS:
Device: miRNA tool — patients to be assessed by the miRNA tool. MicroRNA tool contains miRNA of miR-21、miR-20a-5p、miR-103a-3p、miR-106b-5p、miR-143-5p and miR-215. Investigators evaluate these miRNA status of surgical specimens using qRT-PCR and calculate their risk score(risk score =(0.108×status of miR-21-5p)+(0.086×status of miR-20a-5p)+(0.240×status of miR-103a-3p)+(0.095×status of miR-106b-5p)- (0.238×status of miR-143-5p)-(0.237×status of miR-215),low expression status equals 0 and high expression status equals 1.Then we determine the patients who with a score higher than 1 as exposed patient.

SUMMARY:
The investigators discover the investigators' miRNA tool can be a useful tool to predict the patients with stage II colon who can benefit from chemotherapy.Then the investigators plan to make an observation study that may validation this tool.

DETAILED DESCRIPTION:
This is an observation study. The investigators recruit patients who agree to use their postoperative specimen for miRNA tool examination and receive the investigators' follow up.Their receiving chemotherapy or not will decided by their doctors. The investigators just see whether the stratifying tool could predict prognosis.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent has been obtained from the patient.
* With confirmed diagnosis of stage II colon cancer.
* With moderate/good ECOG health rating (PS): 0-1 score.
* The patient receive no anti-cancer treatment before primary surgery.
* The patient receive radical operation for colon cancer with negative margin.

Exclusion Criteria:

* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.
* Pregnant woman or lactating woman.
* With contraindication to receive adjuvant chemotherapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who had stage II colon cancer and received surgery.They agree to use miRNA tool to test their postoperative specimen.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 years

SECONDARY OUTCOMES:
OS | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wu Song, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- FisrtSunYetsen, Guangzhou, Guangdong, China